CLINICAL TRIAL: NCT04729049
Title: Erector Spinae Plane Block Efficacy Versus Intravenous Morphine for Postoperative Pain Control Following Vertebral Fixation Surgery Via Posterior Approach: a Randomized Controlled Trial
Brief Title: Erector Spinae Block vs Morphine in Vertebral Fixation
Acronym: ATLANTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AUSL Romagna Rimini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1220
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Vertebral Subluxation; Spine Disease; Spondylolisthesis
Keywords: Anesthesia; Postoperative Pain; Postoperative Delirium; Postoperative Nausea and Vomiting; Erector Spine plane Block; Neuraxial anesthesia
MeSH Terms: conditions — Spinal Diseases; Spondylolisthesis; Pain, Postoperative; Emergence Delirium; Postoperative Nausea and Vomiting | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: Cases vs control
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Care provider (anaesthetist) will know the type of anaesthesia performed. Outcome assessor (physician visiting the patient postoperatively) and investigator (study design and data analysis) will not know the type of anaesthesia performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block + patient controlled analgesia (PCA) with intravenous morphine (Experimental): Preoperative bilateral ESP block with ropivacaine 0,4% + dexamethasone 4 mg, 20 mL per side, at the median spinal level of intervention.
  End-surgery: acetaminophen 1 g ev + 4 mg morphine ev before the end of the intervention.
  PCA: morphine 1 mg, max every 30 minutes. Rescue: ketoprofen 100 mg ev, max three times per day.
  Interventions: Procedure: Erector Spinae plane Block; Drug: Patient controlled analgesia with intravenous morphine
- Patient controlled analgesia (PCA) with intravenous morphine (Active Comparator): End-surgery: acetaminophen 1 g ev + 4 mg morphine ev before the end of the intervention.
  PCA: morphine 1 mg, max every 30 minutes. Rescue: ketoprofen 100 mg ev, max three times per day.
  Interventions: Drug: Patient controlled analgesia with intravenous morphine

INTERVENTIONS:
Procedure: Erector Spinae plane Block — Ultrasound-guided interfascial technique, aiming to block the anterior and posterior branches of the spinal nerves for multi-dermatomal analgesia. Injection of local anesthetic in the plane deep to the erector spinae muscles and superficial to the transverse processes, to achieve a craniocaudal distribution along several vertebral levels.
  Other Names: ATLANTE
  Arms: Erector spinae plane block + patient controlled analgesia (PCA) with intravenous morphine
Drug: Patient controlled analgesia with intravenous morphine — Patient-controlled intermittent boluses of morphine 1 mg (maximum once every 15 minutes).
  Other Names: ATLANTE

SUMMARY:
The study aims to shed light about the potential role of Erector Spinae Block in the management of postoperative pain following vertebral fixation surgery via posterior approach. Patients will be randomized, the block will be performed before inducing general anesthesia, intraoperative management will be uniformed, while postoperative analgesia will compare cases (patients who received the block) versus controls (usual care with endovenous morphine infusion only).

DETAILED DESCRIPTION:
The study is a single-centre, interventional, prospective, case-control study. After being informed about the study and potential risks during preoperative anaesthetic evaluation, all patients giving written informed consent will be enrolled in the study.

Inclusion criteria will be: patients undergoing vertebral fixation via posterior approach both for degenerative or traumatic causes, age 18-85, American Society of Anesthesiologists (ASA) I-III, written informed consent signed. Exclusion criteria will be: patients outside the 18-85 year old range, allergies or contraindications to the use of local anaesthetics and erector spinae block, skin infections at the puncture site, body-mass index above 40.

The initial estimate of patients needed to detect statistically significant results has been estimated in 30 (15 cases versus 15 controls). Considering the surgical activity in the organising centre, the study should be completed before the end of 2021. Randomization will be made with a random sequence informatically produced. The study will be double-blinded, with the patient, the nurse doing the postoperative pain assessment and the statisticians not knowing the type of anaesthesia performed (only the anesthesist in the operating theatre is unblinded).

Erector spine plane (ESP) block will be performed after general anaesthesia (GA) induction, with the patient already in prone position. It will be made at the vertebral level of surgical fixation, bilaterally, with Ropivacaine 0.4% and dexamethasone 4 mg in 20 mL of sodium chloride (NaCl) 0.9% per side. GA will be induced with propofol, fentanyl and rocuronium to all patients, while GA maintenance will be performed with total-intravenous anaesthesia (TIVA) with propofol and boluses of fentanyl as required. Basic blood pressure, pulse-oximetry, electrocardiogram, train-of-four, body temperature and bispectral index monitoring will be applied to every patient. At the end of the surgery all the patients will receive a bolus of acetaminophen 1 g and morphine 4 mg.

Post-operative analgesia in controls will be performed by patient-controlled analgesia (PCA) pumps infusing boluses-at-request of morphine 1 mg (maximum once every 15 minutes) with no background infusion, plus acetaminophen 1 g every 8 hours for the first 48 hours.

Post-operative analgesia in cases will be performed with PCA only releasing boluses-at-request (maximum 1 mg every 15 minutes) and acetaminophen 1 g every 8 hours during the first 48 hours.

Postoperative pain will be assessed by a trained physician blinded to the anaesthetic technique employed. Numerical rating scale (NRS) and Richmond agitation-sedation scale (RASS) will be performed at 2-6-12-24-36-48 hours after the end of the surgery.

The primary outcome is postoperative morphine consumption. Secondary outcomes are intraoperative opioid use, postoperative NRS scores, in-hospital length-of-stay and final patient satisfaction.

Statistical analysis will be performed by trained professionals with STATA 14.2 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-III
* written informed consent signed
* traumatic or degenerative disease
* adult age (18-65 year old)

Exclusion Criteria:

* allergies to local anesthetics
* contraindications to ESP block execution
* congenital or drug-induced coagulopathies
* infections at the puncture site
* BMI > 40

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption | 48 hours
  Milligrams of morphine used to control postoperative pain

SECONDARY OUTCOMES:
Intraoperative opioid use | Intraoperative
  Micrograms of fentanyl used to control intraoperative pain
Postoperative pain control | 2-6-12-24-36-48 postoperative hours
  Numeric Rating Scale (NRS) 0= better outcome; 10=worse outcome
Postoperative agitation-sedation-delirium | 2-6-12-24-36-48 postoperative hours
  Richmond agitation-sedation scale RASS -5 Cannot be arouse; 4 Combative
Patients satisfaction | at 48 postoperative hours
  1 (bad) to 10 (good) scale vote
In-hospital length-of-stay | 2-6-12-24-36-48 postoperative hours
  Number of days

CONTACTS AND LOCATIONS:
Overall Officials: Domenico P Santonastaso, MD, Principal Investigator — AUSL Romagna - Ospedale Bufalini di Cesena
Locations (1):
- AUSL Romagna M. Bufalini Hospital, Cesena, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Yes
All data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years, after publication.
Access Criteria: Corresponding author email, upon reasonable request.

REFERENCES:
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] Singh S, Chaudhary NK. Bilateral Ultasound Guided Erector Spinae Plane Block for Postoperative Pain Management in Lumbar Spine Surgery: A Case Series. J Neurosurg Anesthesiol. 2019 Jul;31(3):354. doi: 10.1097/ANA.0000000000000518. No abstract available. PMID 29965831
- [Background] Singh S, Choudhary NK, Lalin D, Verma VK. Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Oct;32(4):330-334. doi: 10.1097/ANA.0000000000000603. PMID 31033625
- [Background] Ueshima H, Inagaki M, Toyone T, Otake H. Efficacy of the Erector Spinae Plane Block for Lumbar Spinal Surgery: A Retrospective Study. Asian Spine J. 2019 Apr;13(2):254-257. doi: 10.31616/asj.2018.0114. Epub 2018 Nov 15. PMID 30424594
- [Derived] Bellantonio D, Bolondi G, Cultrera F, Lofrese G, Mongardi L, Gobbi L, Sica A, Bergamini C, Viola L, Tognu A, Tosatto L, Russo E, Santonastaso DP, Agnoletti V. Erector spinae plane block for perioperative pain management in neurosurgical lower-thoracic and lumbar spinal fusion: a single-centre prospective randomised controlled trial. BMC Anesthesiol. 2023 May 30;23(1):187. doi: 10.1186/s12871-023-02130-z. PMID 37254058